CLINICAL TRIAL: NCT05775575
Title: A Phase Ib/II Study to Investigate the Safety, Tolerance and Pharmacokinetics of TQB3909 With HR-positive, HER2-negative Advanced Breast Cancer
Brief Title: A Clinical Trial of TQB3909 Tablets in Patients With Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-Ib/II-01
Record Dates: First submitted 2022-12-07; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-09

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3909 tablets (Experimental): 200-1000mg of TQB3909 tablets once a day; Oral administration under fast condition, 28 days as a cycle.
  Interventions: Drug: TQB3909 tablets

INTERVENTIONS:
Drug: TQB3909 tablets — TQB3909 is an inhibitor targeting BCL-2 protein

SUMMARY:
TQB3909 is an inhibitor targeting B-cell lymphoma (BCL)-2 protein. By binding to BCL-2 protein, TQB3909 releases Pro apoptotic proteins such as BCL-2-Anatagonist/Killer 1(BAK), BCL-2 associated X (BAX) protein and BCL-2 associated death (BAD) protein, promotes the release of cytochrome c from mitochondria, phosphatidylserine eversion, stimulates caspase 3/7 activity and caspase 3/9 cleavage, and induces apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
* Age: 18 to 75 years old; female patient, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Histopathologically confirmed HR positive and HER2 negative advanced or metastatic breast cancer.
* Patients who have been treated with endocrine therapy and have experienced disease progression.
* Patients previously treated with any CDK4/6 inhibitor and not treated with BCL-2 inhibitor.
* Has at least one measurable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria
* The main organs function well;
* Female patient had no plans to become pregnant and voluntarily took effective contraceptive measures from agree with the study to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* 1. Concomitant disease and medical history:

  1. There were other malignant tumors in 3 years before the first medication.
  2. Has multiple factors affecting oral medication;
  3. Unalleviated toxicity ≥ grade 1 due to any previous therapy;
  4. Major surgical treatment, open biopsy and obvious traumatic injury were performed within 28 days before the study; e．Arteriovenous thrombotic events occurred within 6 months before the first medication, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism; f．Have a history of psychotropic drug abuse and can not quit or have mental disorders; g．Subjects with any severe and / or uncontrolled disease included: Cirrhosis, active hepatitis, history of immunodeficiency;
* Tumor-related symptoms and treatment:

  1. Has central nervous system metastases (CNS) and/or cancerous meningitis or leptomeningeal carcinomatosis;
  2. have received radiotherapy, other antineoplastic therapy within 2 weeks prior to the first dose;
  3. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
* Known hypersensitivity to TQB3909, LHRH agonists (e.g., goserelin), or any excipients.
* Subjects who have received the vaccine within 28 days prior to the first dose, or are planning to receive the vaccine during the study period.
* Has Participated in other clinical trials within 4 weeks before first dose.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patient aged from 18 to 75 years old, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
Enrollment: 65 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (Cycle 1, Day 28)
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred from the first dose to the end of the first treatment cycle.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (Cycle 1, Day 28)
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | Baseline up to 24 months
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3909 tablets in adult patients with Breast cancers

SECONDARY OUTCOMES:
Time to reach maximum (peak)plasma concentration (Tmax) | before administration at Day 1, Cycle1 Day7,Cycle1 Day14, Cycle1 Day28; 1, 2, 4, 6, 8, 10,24,48, and 72 hours after-dose at Day 1; 1, 2, 4, 6, 8, 10, and 24 hours after-dose at Cycle 1 Day 28.
  To characterize the pharmacokinetics of TQB3909 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Peak concentration (Cmax) | before administration at Day 1, Cycle1 Day7,Cycle1 Day14, Cycle1 Day28; 1, 2, 4, 6, 8, 10,24,48, and 72 hours after-dose at Day 1; 1, 2, 4, 6, 8, 10, and 24 hours after-dose at Cycle 1 Day 28.
  Maximum observed concentration (Cmax) of TQB3909
Terminal half-life (T1/2) | before administration at Day 1, Cycle1 Day7,Cycle1 Day14, Cycle1 Day28; 1, 2, 4, 6, 8, 10,24,48, and 72 hours after-dose at Day 1; 1, 2, 4, 6, 8, 10, and 24 hours after-dose at Cycle 1 Day 28.
  Pharmacokinetics parameters to evaluate the half life of TQB3909 (T1/2)
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | before administration at Day 1, Cycle1 Day7,Cycle1 Day14, Cycle1 Day28; 1, 2, 4, 6, 8, 10,24,48, and 72 hours after-dose at Day 1; 1, 2, 4, 6, 8, 10, and 24 hours after-dose at Cycle 1 Day 28.
  To characterize the pharmacokinetics of TQB3909 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) | before administration at Day 1, Cycle1 Day7,Cycle1 Day14, Cycle1 Day28; 1, 2, 4, 6, 8, 10,24,48, and 72 hours after-dose at Day 1; 1, 2, 4, 6, 8, 10, and 24 hours after-dose at Cycle 1 Day 28.
  Cmax,ss is the steady state maximum concentration of TQB3909.
Minimum steady-state plasma drug concentration during a dosage interval (Cmin,ss) | before administration at Day 1, Cycle1 Day7,Cycle1 Day14, Cycle1 Day28; 1, 2, 4, 6, 8, 10,24,48, and 72 hours after-dose at Day 1; 1, 2, 4, 6, 8, 10, and 24 hours after-dose at Cycle 1 Day 28.
  Cmin,ss is the minimum plasma concentration of TQB3909.
Clinilca Benefit Rate (CBR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks.
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Objective Response Rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks.
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No